CLINICAL TRIAL: NCT01062373
Title: Improvement of Polyunsaturated Fatty Acids Status in Premature Newborns Following Docosahexaenoic Acid Enrichment of Human Milk
Brief Title: Effect of Docosahexaenoic Acid (DHA)-Enriched Human Milk in Premature Newborns
Acronym: DHARMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties of recruitement
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C08-20; 2009-A00006-51 (Registry Identifier: IDRCB)
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-01

CONDITIONS: Premature
Keywords: Premature Newborns; Human Milk; DHA; Mother-child
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TG-DHA (Active Comparator): TG-DHA: lactating mothers and their newborn with mothers supplemented with Triglyceride enriched in docosahexaenoic acid
  Interventions: Dietary Supplement: Supplementation of lactating mothers who has delivered prematurely with DHA
- Control (No Intervention): Control: lactating mothers and their newborn with no supplementation given to the mother
- GPL-DHA (Experimental): GPL-DHA: lactating mothers and their newborn with mothers supplemented with Glycerophospholipid enriched in docosahexaenoic acid
  Interventions: Dietary Supplement: Supplementation of lactating mothers who has delivered prematurely with DHA

INTERVENTIONS:
Dietary Supplement: Supplementation of lactating mothers who has delivered prematurely with DHA — Supplementation in DHA will be conducted for 1 month at the dose of 200 mg DHA per day provided by TG-DHA from Decola (products from Martek) (two soft capsules per day)
  Other Names: TG-DHA from Decola compagny in Belgium: oil of microalgae saled by Martek US compagny containing triglycerides enriched in DHA ; code 139 890
  Arms: TG-DHA
Dietary Supplement: Supplementation of lactating mothers who has delivered prematurely with DHA — Supplementation in DHA will be conducted for 1 month at the dose of 200 mg DHA per day provided by GPL-DHA from ASL (10 g per day) (two soft capsules per day)
  Other Names: GPL-DHA from Application Santé des Lipides BioParc Vichy Hauterive France: dry yolk egg powder containing glycerophospholipids enriched in DHA code AA 22/12/11
  Arms: GPL-DHA

SUMMARY:
Several recent publications showed a reduction in the level of DHA and/or an increase in the arachidonic acid (AA)/DHA ratio in the milk of mother. We hypothesized that the polyunsaturated fatty acid (PUFA) status of the premature newborn fed mother's milk is unbalanced because the content of DHA of the milk of mother nowadays is insufficient, whereas scientific arguments point-out the essential role of DHA and balanced AA/DHA ratio of human milk to explain the beneficial role of the breast-feeding at short, medium and long term. We will study the benefits of DHA supplements (TG-DHA versus GPL-DHA) of mothers in PUGA status improvement in their premature newborn consecutive to DHA enrichment and balanced AA/DHA ratio of human milk. GPL-DHA should be more effective than TG-DHA by protecting both n-3 and n-6 fatty acids pathways.

ELIGIBILITY:
Inclusion Criteria:

* Childbirth between 34 and 35 GA
* Breast-feeding
* Caucasian
* Affiliation to social security
* Obtained consent from mother, and parents for the child
* Mother with balanced diet
* No allergy to eggs
* Single pregnancy

Exclusion Criteria:

* Allergy to egg
* Unbalanced diet
* Diabetes
* Known digestive disease
* Counter-indication with breast-feeding
* Cigarettes (more than 5 per day)
* Alcoholism (daily consumption of alcohol)
* Multiple pregnancy

Ages: 1 Day to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To improve PUFA status in premature newborns | 30 days

SECONDARY OUTCOMES:
PUFA in human milk (HM) and mothers | 6 months
Impact on HM bioactives | 6 months
Change in inflammation and oxydative stress | 6 months
Genes expression in newborns | 6 months
Link between mothers genetics and HM DHA level | 6 months
Newborn survey at 6 month-old | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Millet, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Service de Médecine néonatale, Hôpital de la Conception, Marseille, France